CLINICAL TRIAL: NCT07375368
Title: Evaluation of a 3D-Printed Extraoral Camera Assembly for Standardization of Dental Photography:A Randomized Controlled Clinical Trial
Brief Title: Assessment of a 3D-Printed Extraoral Camera Assembly for Standardized Dental Photography
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Adayil, Lecturer, Department of Periodontology Faculty of Dentistry, Cairo University, Cairo University
Other Study IDs: 10.25
Record Dates: First submitted 2026-01-15; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Imaging
Keywords: 3D-printed extraoral camera; standardization; extraoral camera

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study investigates whether a 3D-printed extraoral camera assembly improves the reproducibility and dimensional standardization of dental photographs compared with conventional DSLR photography using standardized settings. The assembly, serving as the index test, standardizes camera position, distance, and angle during image capture, allowing performance comparison with traditional DSLR methods under identical exposure and lighting conditions. By enhancing photographic consistency, the assembly aims to improve longitudinal periodontal records, esthetic documentation, and digital analyses, providing a non-contact, operator-independent tool for reliable visual comparisons across clinical sessions.

ELIGIBILITY:
Inclusion Criteria:

* Adult volunteers aged 18-40 years.
* Intact anterior dentition and healthy periodontal tissues.
* Cooperative and able to maintain a standardized head position. Only intraoral photographs will be taken

Exclusion Criteria:

* Facial deformities or scars affecting the image region.
* Previous orthognathic or periodontal plastic surgery altering soft-tissue contour.
* Active dermatologic lesions or tattoos in the perioral area.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will include adult volunteers aged 18-40 years with intact anterior dentition and healthy periodontal tissues, who are cooperative and able to maintain a standardized head position during imaging. Only intraoral photographs will be captured. Exclusion criteria comprise individuals with facial deformities or scars affecting the photographic region, those who have undergone orthognathic or periodontal plastic surgery altering soft-tissue contours, and participants with active dermatologic lesions or tattoos in the perioral area.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Difference between photographic and actual tooth dimensions (assembly vs standard) | through study completion, an average of 2 weeks